CLINICAL TRIAL: NCT06432777
Title: Recurrent Campylobacter Bacteraemia in Immunocompromised Patients: a Retrospective Nationwide Study in France, 2000-2025
Brief Title: Recurrent Campylobacter Bacteraemia in Immunocompromised Patients
Acronym: CABARET
Status: Not yet recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL24_0512
Record Dates: First submitted 2024-05-14; First posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Campylobacter Infections
Keywords: primary immunodeficiency; Campylobacter; Relapsing bacteraemia
MeSH Terms: conditions — Campylobacter Infections; Primary Immunodeficiency Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Recurrent Campylobacter bacteraemia: Patients presenting at least two distinct episodes of Campylobacter bacteraemia separated by minimum 60 days and an immunodeficiency (innate or acquired)
  and followed by a French hospital
  Interventions: Other: Characteristics of patients and Campylobacter bacteraemia episodes

INTERVENTIONS:
Other: Characteristics of patients and Campylobacter bacteraemia episodes — Variables: characteristics of the patients (demographic characteristics; characteristics of immunodeficiency: diagnosis, immunoglobulin dosage, white cells count etc.; chronic inflammatory bowel disease [IBD]), the bacteria (species, antimicrobial susceptibility) and the infection (clinical presentation, evolution, treatment received)

SUMMARY:
Some rare cases of recurrent Campylobacter bacteraemia (RCB) exist with relapses months to years after an effective treatment and a negativation of all bacterial samples.

As of today, only around 20 cases have been described in the international literature for the last 30 years. The cases are likely highly underreported.

No study describes those recurrent Campylobacter bacteraemias at the scale of a country.

The aim of this multicentre, nationwide, retrospective study is to describe their precise epidemiology in France for the last 25 years, the immune profile of the patients, the specificities of the bacteria involved, the treatments received and the evolution of these infections.

The perspective is to propose a standardization of the medical care of those patients mainly by describing the effective treatments and the explorations of the immune system which should be considered.

ELIGIBILITY:
Inclusion Criteria:

* 2 episodes or more of Campylobacter bacteraemia separated by at least 60 days
* AND immunodeficiency condition
* followed by a French hospital

Exclusion Criteria:

-Opposition of the patient

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: French hospitals
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Description of the characteristics of the patients presenting with recurrent Campylobacter bacteraemia | Baseline
  -demographic characteristics
Description of the characteristics of the patients presenting with recurrent Campylobacter bacteraemia | Baseline
  -characteristics of immunodeficiency: diagnosis, immunoglobulin dosage, white cells count, polyvalent Ig replacement therapy
Description of the characteristics of the patients presenting with recurrent Campylobacter bacteraemia | Baseline
  -chronic inflammatory bowel disease [IBD]
Description of the characteristics of the patients presenting with recurrent Campylobacter bacteraemia | Baseline
  -characteristics of bacteraemia: clinical presentation, bacteria (species, antimicrobial susceptibility), secondary localizations, evolution, treatment modalities (antibiotics and immunother

CONTACTS AND LOCATIONS:
Locations (1):
- Infectious diseases department, Hospital de la Croix Rousse,, Lyon, France

IPD SHARING:
Plan to Share IPD: No